CLINICAL TRIAL: NCT05384665
Title: Impact of Opioids on Heart Rate During Rapid Sequence Intubation: Double-blind Randomized Controlled Study
Brief Title: Impact of Opioids on Heart Rate During Rapid Sequence Intubation
Acronym: CANDY-CRASH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: rate of inclusion too low
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EUCT 2022-500369-28-00
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Rapid Sequence Induction
MeSH Terms: interventions — Remifentanil; Sufentanil

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (placebo + remifentanil) (Experimental)
  Interventions: Drug: Remifentanil; Drug: Placebo
- Group B (sufentanil + placebo) (Experimental)
  Interventions: Drug: Sufentanil; Drug: Placebo
- Group C (placebo + placebo) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Remifentanil — REMIFENTANIL, 5 µg/cc, solution for injection, 0.5 µg/kg, parenteral (intravenous) route, injection delay of 30 seconds, once only
  Arms: Group A (placebo + remifentanil)
Drug: Sufentanil — SUFENTANIL, 5 µg/cc, solution for injection, 0.2 µg/kg, parenteral (intravenous) route, bolus over 5 seconds, once
  Arms: Group B (sufentanil + placebo)
Drug: Placebo — PLACEBO contains 0.9% NaCl, parenteral (intravenous), bolus, one-time

SUMMARY:
The patient is seen upstream by an anaesthetists resuscitator (MAR) in order to carry out his anesthesia consultation. If the patient meets the eligibility criteria he will be informed of the study and his signed consent will be obtained.

Patients will be divided into 3 parallel groups :

* Group A (placebo +remifentanil)
* Group B (sufentanil + placebo)
* Group C (placebo + placebo)

Constants are taken at T0. A non-invasive continuous monitoring (Clearsight ©) will be used to collect data: blood pressure, heart rate, cardiac output.

To ensure double-blinding the nurse who prepares the syringes is not part of the anesthesia team. He/she numbers them in syringe n°1 and n°2 to indicate the order of injection to the MAR.

The MAR injects the drugs according to the standardized study plan (see below):

* T1: the patient receives an intravenous bolus (IV) over 5 seconds of molecule n°1
* 3 minute delay
* Patient receives Etomidate 0.3 mg/kg IV over 10 seconds
* 5 second delay
* The patient receives an IV bolus over 30 seconds of molecule n°2
* 5 second delay
* The patient receives Succinylcholine or Rocuronium IV over 5 seconds
* T2: End of induction, oro-tracheal intubation (= T2)

The laryngoscopy is performed by an experienced MAR or nurse (IADE). The end of the intubation is defined by the fixation of the intubation tube (T3). Hemodynamic parameters are measured every minute for ten minutes after intubation (T4 to T13).

Maintenance of anesthesia is standardized with halogen gas (SEVOFLURANE) and an opioid (SUFENTANIL). Ten minutes after the patient's intubation (T13), the blind is lifted, allowing the addition of sufentanil in groups A and C before any surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 65 years old and any possible ASA OR Patient aged 55 to 65 years old with an ASA ≥ 3,
* Patient undergoing surgery (urgent or scheduled), requiring general anesthesia in rapid sequence, because considered to have a "full stomach", i.e. with: gastro-oesophageal pathology or gastroparesis or a history of bariatric surgery or food intake within two hours for liquids and within six hours for solids,
* Patient informed of the study who gave their written consent before starting the study procedures,
* Patient affiliated to a French social security system.

Exclusion Criteria:

* Patient < 55 years old,
* Patient on beta blockers,
* Atrial fibrillation or other rhythm or conduction disturbances,
* Patient in hemodynamic failure and/or on catecholamines before the start of GA,
* Patient having a history of stroke, hemorrhagic and/or ischemic and/or transient
* Combination with opioid agonists-antagonists or partial opioid antagonists
* Known hypersensitivity to one of the study drugs or to opioids,
* History of difficult intubation,
* Patient under guardianship, curatorship or deprived of liberty,
* Patient participating in another interventional clinical research,
* Patient under AME (State Medical Aid)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
heart rate beats per minute | T2 : oro-tracheal induction
  Absolute variation of heart rate beats per minute between T0 (reference value at the entrance into the operating room) and T2 (end of induction and oro-tracheal intubation)

SECONDARY OUTCOMES:
Cormack score | T2 : oro-tracheal induction
  Cormack score in each group
Laryngoscopy of Macintosh number | T2 : oro-tracheal induction
  Laryngoscopy number for each group
Use of a long bent mandrel | T2 : oro-tracheal induction
  Use of a long bent mandrel for each group
assess side effects according to the opioids used | T2 : oro-tracheal induction
  Percentage of patients with intraoperative vomiting at T2 for each group
assess side effects according to the opioids used | before T2 : oro-tracheal induction
  Percentage of patients requiring vasopressor before T2
assess side effects according to the opioids used | T2 : oro-tracheal induction
  Percentage of patients with thoracic rigidity and/or bradycardia < 50/min at T2 for each group
assess significant variation in hemodynamic responses | T2 : oro-tracheal induction
  Absolute and relative variations of +-20% in SAP/DAP and MAP between T0 and T2
assess significant variation in hemodynamic responses | T13 (10 minutes after intubation)
  Absolute and relative variations of +/- 20% in SAP/DA and MAP between T0 and T13
assess significant variation in hemodynamic responses | T2 : oro-tracheal induction
  Relative variation of +/- 20% of HR between T0 and T2
assess significant variation in hemodynamic responses | T13 (10 minutes after intubation)
  Absolute and relative variations of +/- 20% of HR between T0 and T13.

CONTACTS AND LOCATIONS:
Overall Officials: Marine FONTAINE, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No